CLINICAL TRIAL: NCT05506267
Title: Development of a Tracheal Sound Sensor for Early Detection of Hypoventilation
Brief Title: Development of a Tracheal Sound Sensor
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); RTM Vital Signs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 20C.100; 15294 (Other: Thomas Jefferson University); 1R41DA047779-01 (NIH)
Record Dates: First submitted 2022-08-02; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Insufficiency; Opioid Overdose; Hypoventilation
MeSH Terms: conditions — Respiratory Insufficiency; Opiate Overdose; Hypoventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Trachea Sound Sensor (TSS) — Use the TSS and commercial vital sign monitors to develop a diagnostic algorithm that detects and predicts hypoventilation due to opioids and anesthetic medication

SUMMARY:
An observational study will be conducted in 20 hospitalized surgical patients routinely managed with opioids for anesthesia and post-operative pain control. Trachea Sound Sensor measurements and reference respiratory measurements will be recorded and analyzed to develop diagnostic algorithms that produce a risk-index score that detects/predicts progression from mild hypoventilation, to moderate hypoventilation, to severe hypoventilation due to opioids and other medications that cause respiratory depression.

Our current Trachea Sound Sensor (TSS) has a wired Sony commercial microphone integrated into a commercial pediatric stethoscope, coupled to the skin surface over the trachea at the sternal notch. The Trachea Sound Sensor will measure and record the sounds of air moving within the proximal trachea during inhalation and exhalation. The microphone signal will be converted into an accurate measurement of the patient's respiratory rate and tidal volume (during inhalation & exhalation) over time, to determine the minute ventilation trend, breathing patterns, apnea episodes, and degree of snoring (due to partial upper airway obstruction).

A commercial respiratory facemask and two pneumotachs (gas flow sensors) will also be used to accurately and continuously measure the patient's respiratory rate and tidal volume (during inhalation & exhalation) to determine the minute ventilation trend, breathing patterns, and apnea episodes.

TSS data and reference respiratory data will be collected prior to surgery with the patient breathing normally (baseline), in the Operating Room (OR) during the induction and maintenance of anesthesia, in the Post Anesthesia Care Unit (PACU), and on the general nursing floors of Thomas Jefferson University Hospital (TJUH).

The sounds of air flowing through the proximal trachea will be correlated with the reference breathing measurements using signal processing methods to optimize the measurement accuracy of RR, TV, breathing pattern, apnea episodes, and degree of snoring. A commercial accelerometer may be coupled to the skin surface of the neck (with tape) to measure body position and activity level. The TSS and vital sign trend data will be analyzed to produce a Risk-Index Score every 30 seconds with alerts and alarms that warn the patient and caregivers about progressive Opioid Induced Respiratory Depression (OIRD).

DETAILED DESCRIPTION:
RTM's Trachea Sound Sensor (TSS) and data acquisition system will be used to measure and record the sounds of air movement within the trachea during inhalation/exhalation prior to surgery (baseline), and during management with opioid medications in the operating room (OR), post-anesthesia care unit (PACU), intensive care unit (ICU), and/or general nursing floor.

The TSS will be adhered to the skin of the neck (within the sternal notch) to measure and record the sounds of air flowing through the proximal trachea during inhalation and exhalation. A commercial miniature accelerometer sensor may also be adhered to the skin of the neck and used to measure and record the patient's body position and activity level.

In addition, research staff will intermittently measure and record each patient's respiratory rate (RR) and tidal volume (TV) prior to surgery (baseline), during anesthesia (OR), during anesthesia recovery (PACU), and during post-operative care (ICU or nursing floor) using a commercial research facemask and respiratory flow sensors (pneumotachs) hardwired to a data acquisition system and personnel computer (PC). One commercial pneumotach will accurately measure the patient's tidal volume during inhalation, and another commercial pneumotach will accurately measure the patient's tidal volume during exhalation.

The concentration of oxygen in the inspired air delivered into the facemask will be tightly controlled, according to a physician's order and standard-of-care methods. The facemask and commercial ventilation measurement system was designed and tested in collaboration with Nick Rudolph from the company Hans Rudolph, Inc.

Capnography will also be used to continuously measure and record the concentration of carbon dioxide within the facemask's air during inhalation and exhalation, using end-tidal measurements to estimate the concentration carbon dioxide in the alveoli and arterial blood. Hemoglobin oxygen saturation will be continuously measured and recorded using a commercial pulse oximeter and finger probe.

In some of the study subjects, blood will be intermittently sampled from a radial artery catheter (previously inserted for clinical care) or a peripheral venous catheter and used to measure the levels of pH, oxygen, carbon dioxide, lactate and other analytes using a point-of- care meter. Blood may be sampled more frequently before and after an opioid bolus or a change in opioid dose. Blood will not be sampled from some of the study subjects because a radial artery/venous catheter were not available or functional for blood sample acquisition.

Trend data will be used to develop a diagnostic algorithm with a risk-index score that detects/predicts progression from mild hypoventilation, to moderate hypoventilation, to severe hypoventilation due to opioids

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for inpatient surgery at Thomas Jefferson University Hospital that would routinely receive opioids for their clinical care.
* Age 18 to 80 years.
* Body Mass Index < 35.
* Stable lung function, oxygenation, and ventilation prior to the surgical procedure.
* Stable cardiac, vascular, renal, hepatic, neurologic, gastrointestinal, or muscular function prior to the surgical procedure

Exclusion Criteria:

* Patients scheduled for inpatient surgery at TJUH that would not routinely receive opioids for their clinical care.
* Age < 18 and > 80 years.
* Body Mass Index > 35.
* History of difficult airway management or difficult endotracheal intubation
* History of severe seep apnea, requiring oxygen therapy, or CPAP management at home.
* Unstable pulmonary, cardiac, vascular, renal, hepatic, immune, neurologic, gastrointestinal, or muscular function prior to the surgical procedure.
* Excessive facial hair that may prevent a tight seal around the respiratory facemask.
* Pregnancy
* Patients that decline to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for inpatient surgery at Thomas Jefferson University Hospital that would routinely receive opioids for their clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Develop an algorithm that utilizes the Trachea Sound Sensor sound data to measure respiratory rate with sufficient accuracy for clinical care. | 24 hours
  The wearable Trachea Sound Sensor (TSS) will measure and analyze the sounds of air flow in the trachea during inhalation and exhalation to calculate respiratory rate (RR). Calibrated pneumotachs attached to a tight fitting face mask and a capnometer will be used to simultaneously measure the patient's RR. TSS measurements and reference respiratory measurements will be analyzed and correlated using a transfer function algorithm to calculate respiratory rate with sufficient accuracy for clinical care (+/- 1 breath per minute accuracy)
Develop an algorithm that utilizes the Trachea Sound Sensor sound data to measure tidal volume (TV) with sufficient accuracy for clinical care. | 24 hours
  The wearable Trachea Sound Sensor (TSS) will measure and analyze the sounds of air flow in the trachea during inhalation and exhalation to calculate tidal volume (TV). Calibrated pneumotachs attached to a tight fitting face mask will be used to simultaneously measure the patient's TV. TSS measurements and reference respiratory measurements will be analyzed and correlated using a transfer function algorithm to calculate an approximate tidal volume with sufficient accuracy for clinical care (+/- 100 milliliters per breath accuracy)
Develop an algorithm that utilizes the Trachea Sound Sensor sound data to measure tidal volume (TV) with sufficient accuracy for clinical care. | 24 hours
  The wearable Trachea Sound Sensor (TSS) will measure and analyze the sounds of air flow in the trachea during inhalation and exhalation to calculate tidal volume (TV). Calibrated pneumotachs attached to a tight fitting face mask will be used to simultaneously measure the patient's TV. TSS measurements and reference respiratory measurements will be analyzed and correlated using a transfer function algorithm to calculate tidal volume with sufficient accuracy for clinical care. TSS measurements of TV will be categorized into one of five bands (normal TV, decreased TV, very decreased TV, increased TV, very increased TV) with 95% accuracy.
Develop an algorithm that utilizes the Trachea Sound Sensor sound data to measure the duration of apnea with sufficient accuracy for clinical care. | 24 hours
  The wearable Trachea Sound Sensor (TSS) will measure and analyze the sounds of air flow in the trachea during inhalation and exhalation to calculate duration of apnea (seconds). Calibrated pneumotachs attached to a tight fitting face mask and a capnometer will be used to simultaneously measure the duration of apnea. TSS measurements and reference respiratory measurements will be analyzed and correlated using a transfer function algorithm to calculate the duration of apnea (10 to 15 seconds, 16 to 30 seconds, > 30 seconds) with 95% accuracy.
Development of a Diagnostic Algorithm with a Risk-Index Score that Detects and Predicts Hypoventilation due to Opioids and Anesthetic Medications | 24 hours
  A wearable Trachea Sound Sensor (TSS) will measure and analyze the sounds of air flow in the trachea during inhalation and exhalation to calculate RR, TV, and duration of apnea. A commercial pulse oximeter will simultaneously measure heart rate and hemoglobin oxygen saturation. A commercial capnometer will simultaneously measure respiratory rate, duration of apnea, and end-tidal carbon dioxide concentration. The TSS measurements and reference respiratory measurements will be recorded and analyzed to develop a diagnostic algorithm with a risk index score (RIS) that detects/predicts the progression from normal ventilation to hypoventilation due to opioids and other medications that cause respiratory depression. The TSS and vital sign trend data will be analyzed to produce a Risk-Index Score updated every 30 seconds with alerts that warn the patient and caregivers about progressive Opioid Induced Respiratory Depression (OIRD) with > 90% sensitivity and specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen McNulty, DO, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadollahi A, Moussavi ZM. Acoustical respiratory flow. A review of reliable methods for measuring air flow. IEEE Eng Med Biol Mag. 2007 Jan-Feb;26(1):56-61. doi: 10.1109/memb.2007.289122. No abstract available. PMID 17278773
- [Background] Volkow ND, Collins FS. The Role of Science in the Opioid Crisis. N Engl J Med. 2017 Nov 2;377(18):1798. doi: 10.1056/NEJMc1711494. No abstract available. PMID 29117474
- [Background] Yu L, Ting CK, Hill BE, Orr JA, Brewer LM, Johnson KB, Egan TD, Westenskow DR. Using the entropy of tracheal sounds to detect apnea during sedation in healthy nonobese volunteers. Anesthesiology. 2013 Jun;118(6):1341-9. doi: 10.1097/ALN.0b013e318289bb30. PMID 23407106
- [Background] Ramsay MA, Usman M, Lagow E, Mendoza M, Untalan E, De Vol E. The accuracy, precision and reliability of measuring ventilatory rate and detecting ventilatory pause by rainbow acoustic monitoring and capnometry. Anesth Analg. 2013 Jul;117(1):69-75. doi: 10.1213/ANE.0b013e318290c798. Epub 2013 Apr 30. PMID 23632055
- [Background] Mildh LH, Scheinin H, Kirvela OA. The concentration-effect relationship of the respiratory depressant effects of alfentanil and fentanyl. Anesth Analg. 2001 Oct;93(4):939-46. doi: 10.1097/00000539-200110000-00028. PMID 11574361
- [Background] Shafer SL, Varvel JR, Aziz N, Scott JC. Pharmacokinetics of fentanyl administered by computer-controlled infusion pump. Anesthesiology. 1990 Dec;73(6):1091-102. doi: 10.1097/00000542-199012000-00005. PMID 2248388
- [Background] Chen G, de la Cruz I, Rodriguez-Villegas E. Automatic lung tidal volumes estimation from tracheal sounds. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:1497-500. doi: 10.1109/EMBC.2014.6943885. PMID 25570253